CLINICAL TRIAL: NCT05198869
Title: SpotLight-19 Research and Development Study
Brief Title: SpotLight-19 Research & Development Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: ISBRG Corp (Other)
Responsible Party: Principal Investigator, Alan Forster, Principal Investigator, Ottawa Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20210902
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spectral scan (All participants) (Other): 1. Fitzpatrick skin assessment.
  2. Fingertip scanned using the SpotLight-19 device. The scan is approximately 10-20 seconds. Participants will not feel any sensation from the device, i.e., no heat, no pain, no cold, no vibration or pressure.
  3. Information collected from the medical record regarding participant age, COVID-19 vaccination status, presence of COVID-19 symptoms, and PCR test result.
  Interventions: Device: Spectral scan

INTERVENTIONS:
Device: Spectral scan — Consenting participants will have a SpotLight-19 scan

SUMMARY:
In this study, we will use the SpotLight-19 device in patients presenting to a coronavirus disease (COVID-19) Assessment Centre for polymerase chain reaction (PCR) testing. Consenting patients will undergo a Spotlight-19 scan. We will link the scan to PCR results, age, vaccination status, and COVID-19 symptoms in order to calibrate the SpotLight-19 prediction algorithm of a state of COVID-19 infection.

DETAILED DESCRIPTION:
Implementation of rapid, accessible, and accurate COVID-19 testing is a cornerstone of public health efforts to contain and respond to the spreading virus. To respond to this need, ISBRG Corp is applying its SpotLight-19 device to the challenge of developing a non-invasive screening test for COVID-19. The SpotLight-19 device is designed to use non-invasive visible and near-infrared (NIR) spectroscopic measurements of an individual's fingertip and an artificial intelligence technology platform calibrated using viral diagnostic measurements to identify and recognize a spectral fingerprint specific to COVID-19.

All individuals (3yrs or older) presenting to designated hospital COVID-19 Assessment Centres in Ottawa will be recruited to participate. Only people with extreme fingertip scarring will be excluded. Consenting participants will undergo a scan using the SpotLight-19 device - this includes a Fitzpatrick Skin Assessment and 10-20 second scans of the fingertip with the SpotLight-19 device. Following the scan participants will undergo a PCR test as per usual care. The PCR result, participant age, COVID-19 vaccination status, and presence of COVID-19 symptoms will be collected from the medical record and shared with ISBRG Corp. A minimum of 250 COVID-19 positive and a minimum of 250 COVID-19 negative as determined by PCR will be sought. The number of enrolled participants to achieve the sample size will depend on the COVID-19 positivity rate.

ELIGIBILITY:
Inclusion Criteria:

* Qualifies for COVID-19 testing as per Assessment Site protocol; or
* Is capable of cooperating with testing
* Is clinically stable such that the testing protocol may be completed safely

Exclusion Criteria:

* Extreme fingertip scarring or other physical condition that prevents use of the device

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12500 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
spectra indicative of COVID-19 infection | immediate upon scan
  specific wavelengths of light that correlate with COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Rae Lake, MD, Principal Investigator — ISBRG Corp
Locations (2):
- Canada (2):
  - COVID-19 CHEO Assessment Centre, Ottawa, Ontario
  - COVID-19 Assessment Centre for Adults, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No